CLINICAL TRIAL: NCT03915171
Title: Sensitivity and Specificity of NGS in Detecting bMSI in Patients With Gastric, Duodenal and Small Intestinal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RSTL2018011
Record Dates: First submitted 2019-03-25; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Gastrointestinal Cancer
Keywords: NGS bMSI Gastrointestinal
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSI-H (Experimental): IHC/PCR tested as dMMR/ MSI-H
  Interventions: Diagnostic Test: Next generation sequencing
- MSS (Experimental): IHC/PCR tested as pMMR/ MSS
  Interventions: Diagnostic Test: Next generation sequencing

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — NGS can provide genetic and MSI test for patients

SUMMARY:
To study the sensitivity and specificity of NGS in detecting Microsatellite State in blood and to evaluate its potential application in gastrointestinal cancer.

DETAILED DESCRIPTION:
NGS can not only detect tissue samples, but also blood samples. For some inoperable cancer patients, the acquisition of tissue samples is difficult and traumatic. It is of great significance for the diagnosis and treatment of these patients to determine MSI status by blood testing. In addition, the heterogeneity of malignant tumors is usually strong, blood testing can overcome the heterogeneity of tissue, and can dynamically monitor the patient's condition. 50 patients with gastric cancer, duodenal cancer and small intestinal cancer will be enrolled in the study. Among them, 30 patients with MSI-H and 20 patients with MSS confirmed by IHC/PCR.The investigators will use 520 gene panel for NGS sequencing of tissue and blood samples from selected patients to study the sensitivity and specificity of NGS in detecting Microsatellite State in blood.

ELIGIBILITY:
Inclusion Criteria:

* Age (>18 years old).
* Histologically diagnosed as gastric cancer, duodenal cancer or small intestinal cancer (stage III, stage IV).
* The status of dMMR/pMMR was confirmed by IHC/PCR.
* with tissue and blood samples (including ctDNA and white blood cells) that meet the requirements.
* Agree to provide demographic, medical history, pathological diagnosis, imaging diagnosis, TNM staging, ECOG score and other information.

Exclusion Criteria:

* Suffering from other malignant tumors at the same time.
* Others that the investigator consider that is inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of blood MSI detected by NGS | 1 year
  To study the sensitivity and specificity of blood MSI detected by NGS.

SECONDARY OUTCOMES:
Ideal sequencing depth of MSI in blood test | 1 year
  To study the ideal sequencing depth of MSI in blood test.
Correlation between MSI status and TMB | 1 year
  To study the correlation between MSI status and TMB.
Correlation between MMR gene and other gene mutations | 1 year
  To study thecorrelation between MMR gene and other gene mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China